CLINICAL TRIAL: NCT05573893
Title: Prospective Non-interventional Study (NIS) to Examine Patient-reported Outcomes and Real-world Clinical Data in Patients With HER2-positive, HER2-low or HER2-ultralow Unresectable or Metastatic Breast Cancer Treated With Trastuzumab Deruxtecan
Brief Title: PROVIDENCE - Prospective Non-interventional Study (NIS) to Examine Patient-reported Outcomes and Real-world Clinical Data in Patients With HER2-positive, HER2-low or HER2-ultralow Unresectable or Metastatic Breast Cancer Treated With Trastuzumab Deruxtecan
Acronym: PROVIDENCE
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00028
Record Dates: First submitted 2022-09-29; First posted 2022-10-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms; Breast Cancer; Neoplasm Metastasis
Keywords: Trastuzumab-Deruxtecan,; Human epidermal growth factor receptor 2 Positive Breast Cancer,; Human epidermal growth factor receptor 2 Low Breast Cancer,; Human epidermal growth factor receptor 2 Ultralow Breast Cancer,
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 containing patients with documented HER2-positive unresectable or metastatic BC receiving T-DXd treatment in line with the applicable summary of product characteristics (SmPC) within routine clinical practice.
- Cohort 2: Cohort 2 containing patients with documented HER2-low or HER2-ultralow unresectable or metastatic BC receiving T-DXd treatment in line with the applicable summary of product characteristics (SmPC) within routine clinical practice.

SUMMARY:
This is a prospective non-interventional, multicenter study observing patient reported outcomes as well as real-world efficacy and safety of trastuzumab deruxtecan (T-DXd) in patients with documented Human epidermal growth factor receptor 2 (HER2)-positive, HER2-low or HER2-ultralow unresectable or metastatic breast cancer (BC) receiving T-DXd in line with the applicable summary of product characteristics (SmPC) within routine clinical practice in Germany. In addition, patients will be informed about use of digital healthcare application (DiGA).

DETAILED DESCRIPTION:
Eligible participants will be those patients with documented HER2-positive, HER2-low or HER2-ultralow unresectable or metastatic BC receiving T-DXd treatment in line with the applicable summary of product characteristics (SmPC) within routine clinical practice.

All diagnostic and treatment procedures including visit frequency are at the discretion of the treating physician and not defined by the protocol. T-DXd treatment is considered as a selection criteria. Patients will be informed about use of digital healthcare application (DiGA).

Approximately 800 eligible participants will be enrolled which includes 400 patients in the HER2-positive cohort and 400 patients in the HER2-low/ HER2-ultralow cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old
2. Patients (irrespective of sex and gender) with pathologically documented breast cancer that:

   * is unresectable or metastatic
   * has confirmed HER2+, HER2-low or HER2-ultralow tumor status by local pathology
   * was previously treated with one or more anti-HER2 directed therapy if the tumor is HER2+ OR
   * was previously treated with at least one endocrine therapy in the metastatic setting and is not considered suitable for endocrine therapy as the next line of treatment if the tumor is HR+, HER2-low or HER2-ultralow OR
   * was previously treated with prior chemotherapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy if the tumor is HER2-low.
3. Has documented radiologic progression (during or after most recent treatment)
4. Patient is eligible for T-DXd treatment in line with the specifications mentioned in the ENHERTU® SmPC and is scheduled for T-DXd treatment *
5. Patient is able to read and understand either German or English
6. Signed written informed consent

   * The prescription of the medicinal product is clearly separated from the decision to include the patient in this NIS.

Exclusion Criteria:

1. Start of T-DXd treatment for more than 30 days before enrolment (eCRF registration date)
2. Known hypersensitivity to T-DXd or any of the excipients of the drug
3. Pregnancy or breast feeding
4. Current or planned participation in an interventional clinical trial
5. Current or planned systemic treatment of any tumor other than unresectable or metastatic BC

Patients who have never received any T-DXd dose will be discontinued from the study and will be considered as a late screening failure, no further documentation besides reason and date of discontinuation is needed.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented Human epidermal growth factor receptor 2 (HER2)-positive, HER2-low or HER2-ultralow unresectable or metastatic breast cancer (BC) receiving T-DXd in line with the applicable summary of product characteristics (SmPC) within routine clinical practice may participate in this NIS.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-world Time To Next Treatment (rwTTNT1) | From first dose of T-DXd until initiation of subsequent therapy or death of any cause, whichever came first, assessed up to 60 months
  rwTTNT1 is defined as the time from T-DXd initiation to initiation of subsequent therapy

SECONDARY OUTCOMES:
Change in HRQoL based on FACT-B questionnaire at 6 months after baseline | 6 months
  To evaluate patient-reported outcomes (PROs)/ health-related quality of life (HRQoL) based on FACT-B questionnaire at 6 months after baseline. The Functional Assessment of Cancer Therapy - Breast (FACT-B) is a 37-item instrument designed to measure five domains of HRQoL in breast cancer patients: Physical, social, emotional, functional well-being as well as a breast-cancer subscale (BCS). FACT-B will be collected electronically at time points synchronized with clinic visits during the study.
Change in HRQoL based on FACT-G questionnaire at 6 months after baseline | 6 months
  To evaluate patient-reported outcomes (PROs)/ health-related quality of life (HRQoL) based on FACT-G questionnaire at 6 months after baseline. The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of HRQoL in cancer patients: Physical, social, emotional, and functional well-being. FACT-G will be collected electronically at time points synchronized with clinic visits during the study.

OTHER OUTCOMES:
Change in HRQoL based on FACT-B questionnaire compared to baseline over time | Patient questionnaires will be collected at time points synchronised with clinic visits during study, assessed up to 60 months
  Defined as changes in FACT-B (total score and subscale domains) at different timepoints compared to baseline. The Functional Assessment of Cancer Therapy - Breast (FACT-B) is a 37-item instrument designed to measure five domains of HRQoL in breast cancer patients: Physical, social, emotional, functional well-being as well as a breast-cancer subscale (BCS).
Change in HRQoL based on EQ-5D questionnaire compared to baseline over time | Patient questionnaires will be collected at time points synchronised with clinic visits during study, assessed up to 60 months
  Defined as changes in EQ-5D (subscale domains and VAS) at different timepoints compared to baseline.
  EQ-5D is a standardized instrument for use as a measure of patient-reported health outcomes (Euro-QoL). The 5 health-state dimensions in the EQ-5D-5L include: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-point scale from 1 (no problem) to 5 (unable to/extreme problems). The EQ-5D-5L also includes a graded (0 to 100) vertical visual analog scale (EQ VAS) on which the participant rates his or her general state of health at the time of the assessment.
Real-world Overall Response Rate (rwORR) | From first dose of T-DXd until end of T-DXd treatment or death of any cause, whichever came first (investigator-assessed according to clinical routine), assessed up to 60 months
  rwORR is defined as percentage of patients having complete response or partial response as best response as determined by the investigator
Real-world Progression-free Survival (rwPFS) | From first dose of T-DXd until disease progression (investigator-assessed according to clinical routine) or death of any cause, whichever came first, assessed up to 60 months
  rwPFS is defined as time from T-DXd initiation to the date of the first source evidence for progression referenced by the clinician (e. g., radiology/ pathology report date) or the date of clinician note when no other corresponding evidence sources were documented) or death, whichever occurs first
Real-world Overall Survival (rwOS) | From first dose of T-DXd until death of any cause, assessed up to 60 months
  rwOS is defined as time from T-DXd initiation to date of death
Real-world Time To Treatment Discontinuation (rwTTD) | From first dose of T-DXd until discontinuation of T-DXd treatment therapy or death of any cause, whichever came first, assessed up to 60 months
  rwTTD is defined as time from T-DXd initiation to discontinuation, or death
Real-world Time To Next Treatment 2 (rwTTNT2) | From first dose of T-DXd until initiation of second subsequent therapy or death of any cause, whichever came first, assessed up to 60 months
  rwTTNT2 is defined as time from initiation of T-DXd treatment to initiation of second next treatment, or death
Real-world Time to Treament Discontinuation 2 (rwTTD2) | From first dose of T-DXd until discontinuation of corresponding subsequent therapy or death of any cause, whichever came first, assessed up to 60 months
  rwTTD2 is defined as time from initiation T-DXd treatment to discontinuation of corresponding subsequent therapy, or death
Real-world Progression-free Survival (rwPFS2) | From first dose of T-DXd until second disease progression (investigator-assessed according to clinical routine) or death of any cause, whichever came first, assessed up to 60 months
  rwPFS2 is defined as time from T-DXd initiation to the date of the first source evidence for the second progression referenced by the clinician (e. g., radiology/ pathology report date) or the date of clinician note when no other corresponding evidence sources were documented) or death, whichever occurs first
Safety: Collection of Adverse Events (AE) | during routine visits, up to 60 months
  Safety evaluated based on type of Adverse Event (AE), intensity, causal relationship to treatment, duration, handling, outcome, and seriousness
T-DXd dose modifications | during routine visits, up to 60 months
  To evaluate treatment modifications in patients treated with T-DXd in a real-world setting
Description of DiGA user and non-user population | assessed up to 60 months
  Age, Education, Family status, depressive mood, diagnostic testing, HR-status, Stage IV at initial diagnosis, localization of metastases, presence or history of (in) active brain metastases, previous therapies, subsequent therapies, center characteristics, DiGA usage

CONTACTS AND LOCATIONS:
Locations (94):
- Germany (94):
  - Research Site, Amberg
  - Research Site, Ansbach
  - Research Site, Apolda
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bad Reichenhall
  - Research Site, Baden-Baden
  - Research Site, Balingen
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bonn
  - Research Site, Brandenburg
  - Research Site, Braunschweig
  - Research Site, Bremen
  - Research Site, Bremerhaven
  - Research Site, Coburg
  - Research Site, Dessau
  - Research Site, Donauwörth
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Eggenfelden
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Filderstadt - Bonlanden
  - Research Site, Frankfurt
  - Research Site, Freudenstadt
  - Research Site, Fürstenfeldbruck
  - Research Site, Fürstenwalde
  - Research Site, Gerlingen
  - Research Site, Giessen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidenheim
  - Research Site, Heilbronn
  - Research Site, Hildesheim
  - Research Site, Homburg/Saar
  - Research Site, Jena
  - Research Site, Kaiserslautern
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kempten
  - Research Site, Kiel
  - Research Site, Kulmbach
  - Research Site, Landshut
  - Research Site, Leer
  - Research Site, Leipzig
  - Research Site, Loerrach
  - Research Site, Lübeck
  - Research Site, Lüneburg
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Memmingen
  - Research Site, Mönchengladbach
  - Research Site, Mutlangen
  - Research Site, Mühlhausen
  - Research Site, München
  - Research Site, Neumarkt
  - Research Site, Neustadt am Rübenberge
  - Research Site, Nordhausen
  - Research Site, Nuremberg
  - Research Site, Oldenburg
  - Research Site, Oranienburg
  - Research Site, Potsdam
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Rosenheim
  - Research Site, Rotenburg (Wümme)
  - Research Site, Saalfeld
  - Research Site, Saarbrücken
  - Research Site, Salzwedel
  - Research Site, Schwäbisch Hall
  - Research Site, Siegen
  - Research Site, Singen
  - Research Site, Solingen
  - Research Site, Stade
  - Research Site, Stuttgart
  - Research Site, Torgau
  - Research Site, Troisdorf
  - Research Site, Ulm
  - Research Site, Walsrode
  - Research Site, Weiden
  - Research Site, Weinheim
  - Research Site, Weisenfels
  - Research Site, Westerstede
  - Research Site, Wiesbaden
  - Research Site, Winnenden
  - Research Site, Wolfsburg
  - Research Site, Wuppertal
  - Research Site, Würzburg
  - Research Site, Zittau

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home